CLINICAL TRIAL: NCT01150006
Title: Correlation Between Various Adipokines and Vascular Inflammation Measured by 18FDG-PET In Healthy Male Subjects
Brief Title: Correlation Between Various Adipokines and Vascular Inflammation Measured by Positron Emission Tomography (PET) With 18F-fluoro-deoxyglucose (FDG) (18FDG-PET)
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Name/Official Title: Kyung Mook Choi, Korea University
Other Study IDs: PET_Adipokines
Record Dates: First submitted 2010-06-09; First posted 2010-06-24 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-04

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; vascular inflammation; adipocyte fatty acid binding protein; adiponectin; leptin; 18FDG-PET
MeSH Terms: conditions — Atherosclerosis | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, plasma, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy male participants
  Interventions: Other: Cross sectional study

INTERVENTIONS:
Other: Cross sectional study — This is not intervention study. The purpose of the study is to examine the relationship between various adipokine levels and PET imaging at the cross section setting

SUMMARY:
The inflammatory state and composition of atherosclerotic plaques are considered the main contributing factors responsible for acute cardiovascular events, rather than the degree of stenosis. Recently, positron emission tomography (PET) with 18F-fluoro-deoxyglucose (FDG) has been suggested as a promising novel imaging technique to identify the inflammatory state of atherosclerotic plaque. Recently, a few clinical studies showed that circulating A-FABP level had a close relation with the development of atherosclerosis in human. Therefore, in the present study, the investigators examined the relationship between circulating A-FABP and vascular inflammation of carotid arteries measured using FDG-PET in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers for visiting routine medical check in our clinic

Exclusion Criteria:

* History of cardiovascular disease (myocardial infarction, unstable angina,stroke, or cardiovascular revascularization)
* Diabetes
* Hypertension
* Malignancy
* Severe renal or hepatic disease
* Subjects taking medications that might affect inflammation such as NSIAD and statin

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male participats who underwent a medical health check in the health promotion center in Korea Guro University
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Vascular inflammation in carotid arterial wall, represented as the target-to-background ratio (TBR), using FDG-PET | 12 weeks

SECONDARY OUTCOMES:
Circulating serum A-FABP levels | 12 weeks
Circulating serum leptin levels | 12weeks
Circulating serum adiponectin levels | 12 weeks
Carotid intima-media thickness levels measured using ultrasonography | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mook Choi, MD.PhD, Principal Investigator — Korea University
Locations (1):
- Hye Jin Yoo, Seoul, South Korea